CLINICAL TRIAL: NCT07361315
Title: Development and Online Evaluation of an Online Course for Parasomnias
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Nora Vincent, Psychologist, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS26738
Record Dates: First submitted 2025-11-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Sleep Terror; Sleepwalking; Nightmare Disorder; REM Sleep Behavior Disorder (iRBD); Confusional Arousal
Keywords: Parasomnia course evaluation; online parasomnia
MeSH Terms: conditions — Night Terrors; Somnambulism; REM Sleep Behavior Disorder; Sleep Arousal Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep hygiene control (Active Comparator): Sleep Hygiene Education
  Interventions: Behavioral: Sleep Hygiene Control
- Parasomnia Education (Experimental): Parasomnia Education
  Interventions: Behavioral: Parasomnia Education

INTERVENTIONS:
Behavioral: Parasomnia Education — Week 1: education about types of parasomnias and their causes Week 2: safety planning, relaxation training and imagery rehearsal therapy Week 3: Lucid dreaming, imagery rehearsal therapy, scheduled awakenings Week 4: cognitive therapy, review
  Arms: Parasomnia Education
Behavioral: Sleep Hygiene Control — Week 1: safety planning Week 2: caffeine, cannabis, alcohol, nicotine Week 3: exercising, napping, eating before bed Week 4: noise, light, temperature
  Arms: Sleep hygiene control

SUMMARY:
Parasomnias are unwanted events during sleep. These refer to sleep terrors, sleepwalking, sleep eating, nightmares, and movement during REM sleep. There are few systematic behavioral treatments for these problems and individuals with them often receive little education about self-management. This research examines and evaluates the effectiveness of a 4 week online course providing education and guidance about managing parasomnias. The primary outcomes are improvement in parasomnia frequency and distress. The secondary outcomes are improvements in work and social adjustment, mood, anxiety, stress level, fatigue, sleepiness, insomnia, and cognitive interference.

DETAILED DESCRIPTION:
Parasomnia disorders are prevalent and impactful conditions, however, there are challenges with disseminating evidence-based interventions for these problems. The rationale for this project is to deliver an online evidence-based course for parasomnias to adults with these disorders to provide education and help for these conditions. The objectives are to determine whether participation in the course reduces the frequency and severity of parasomnias, as evaluated using a sleep diary. Study hypotheses are as follows: a) those receiving the course compared to sleep hygiene education will have a reduction in frequency and severity of parasomnias; b) those receiving the online course compared to sleep hygiene education will have a reduction in sleepiness, fatigue, insomnia, perceived cognitive interference, depression, anxiety, stress, and work and social life interference.

This is a single-blind, randomized controlled trial with two conditions (online course, sleep hygiene education). Participants will be 20 adult outpatients referred to the Behavioral Sleep Medicine Clinic at the Health Sciences Center for treatment of a parasomnia.

Participants will be recruited off the waiting list of an outpatient Behavioral Sleep Medicine Clinic. A research coordinator will screen eligible participants over the telephone and obtain informed consent. Following this, participants will be given a study ID# and link to a pre-treatment survey. Once survey materials have been submitted, participants will be randomized to the online course or to weekly sleep hygiene newsletter, through an automated randomization service. Both groups will monitor their sleep throughout the study using a sleep diary (daily), and complete several questionnaires (weekly). The online course will consist of 4 weekly virtual logins and review of material. The control group will consist of receipt of weekly sleep hygiene tips communicated through a newsletter. At the end of 4 weeks, and at a 2 month follow-up, the surveys will be re-administered.

ELIGIBILITY:
Inclusion Criteria:

* physician referred for parasomnia
* meet criteria for parasomnia on the Structured Clinical Interview for Sleep Disorders (SCISD-R)
* age >= 18 years
* parasomnia duration >= 6 months
* English reading, sighted
* access to device.

Exclusion Criteria:

* currently taking one of Lithium, Thioridazine, Chlorpromazine, Perphenazine, Methaqualone, Amitriptyline, Selective Serotonin Re-Uptake Inhibitors, Serotonin and Norepinephrine Re-Uptake inhibitors, or Zopiclone
* seizure or major neurological disorder
* untreated sleep apnea, restless legs syndrome, or narcolepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
self-reported parasomnia severity | baseline, week 4, week 6
  sleep diary recorded parasomnia severity rating (from 0 to 3, with 3 being most severe)
self-reported parasomnia frequency | baseline, week 4, week 6
  frequency of parasomnia events per week (0 to 100)

SECONDARY OUTCOMES:
Secondary measures | baseline, week 4, week 6
  general fatigue (Multi-Dimensional Fatigue Inventory, General Fatigue subscale); scores range from 4 (low fatigue) to 20 (high fatigue)
Sleepiness | baseline, week 4, week 6
  Epworth Sleepiness Scale; scores range from 0 (low sleepiness) to 24 (high sleepiness)
Insomnia Severity | baseline, week 4, week 6
  Insomnia Severity Index; scores range from 0 (absent) to 21 (high)
NREM parasomnia symptoms | baseline, week 4, week 6
  Paris Arousal Disorders Severity Scale; scores range from 0 (absent or low severity) to 50 (high severity)
REM parasomnia symptoms | baseline, week 4, week 6
  REM Sleep Behavior Questionnaire; scores range from 0 (absent or few symptoms) to 13 (more symptoms)
nightmare frequency and severity | baseline, week 4, week 6
  Nightmare Experience Scale; scores range from 0 (absent or less frequent/severe nightmares) to 16 (more frequent/severe nightmares)
Daytime consequences of parasomnias | baseline, week 4, week 6
  Parasomnia Effects Scale; scores range from 0 (less or no consequences) to 120 (more consequences)
Work and Social Interference | baseline, week 4, week 6
  Work and Social Adjustment Scale; scores range from 0 (no interference) to 40 (significant interference)
Perceived Cognition | baseline, week 4, week 6
  PROMIS-Applied Cognition Scale; scores range from 4 (low or no problems with cognition) to 20 (significant problems with cognition)
Mental Health Symptoms | baseline, week 4, week 6
  Depression, Anxiety, and Stress Scale; depression subscale ranges from 0 (low) to 21 (high); anxiety subscale ranges from 0 (low) to 21 (high), stress subscale ranges from 0 (low) to 21 (high)

CONTACTS AND LOCATIONS:
Overall Officials: Norah Vincent, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Psychealth Center, University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
anonymized data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2026-December 2027
Access Criteria: Access upon request to PI (study protocol, informed consent letter, statistical analysis plan